CLINICAL TRIAL: NCT00686413
Title: An Open Label Positron Emission Tomography (PET) Study Using 2-[18F]-F-A85380 to Determine α4β2 Neuronal Nicotinic Receptor Occupancy of AZD3480 After Oral Administration to Healthy Male Subjects (Non Nicotine Users)
Brief Title: Positron Emission Tomography Study Using 2-[18F]-F-A85380 to Determine α4β2 Neuronal Nicotinic Receptor Occupancy of AZD3480 After Oral Administration to Healthy Male Subjects
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans-Göran Hårdemark, MD, PhD, Medical Science Director Clinical Neuroscience TA, AstraZeneca R&D Södertälje
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3690C00018; EudraCT No. 2007-004852-35
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
Keywords: PET; AZD3480; PET examination
MeSH Terms: interventions — ispronicline; 2-fluoro-3-(2-azetidinylmethoxy)pyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD3480
- 2 (Experimental)
  Interventions: Radiation: 2-[18F]-F-A85380

INTERVENTIONS:
Drug: AZD3480 — single dose, oral
  Arms: 1
Radiation: 2-[18F]-F-A85380 — Single dose, IV
  Arms: 2

SUMMARY:
The study is being performed in order to learn more about AZD3480 (potential as treatment for patients with Alzheimer's Disease) and to investigate how much of AZD3480 is bound to the nicotinic receptors in the brain at different concentrations of AZD3480 in blood, as well as to investigate the period of time for this binding.

ELIGIBILITY:
Inclusion Criteria:

* Physically Healthy volunteers
* Genotyped with regard to CYP2D6
* Normal MRI scan at Visit 2

Exclusion Criteria:

* Known or suspected drug or alcohol abuse or positive drugs of abuse screen as judged by the investigator.
* Participation in a PET examination as part of a scientific study during the past twelve months.
* Prescribed or non-prescribed from two weeks prior to the first PET examination. Occasional paracetamol and nasal spray for congestion will be allowed as medication.

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration (AUC, Cmax, tmax) | During time period of the PET assessement
The whole brain uptake and regional distribution of radioligand 2-[18F]-F-A85380 following single intravenous (iv) microdose will be assessed (using derived radioactivity measurements). | One on baseline day and one at the drug treatment day

SECONDARY OUTCOMES:
SafetyAEs and vital signs. | During the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Göran, Hårdemark, MD, PhD, Study Director — Clinical Neuroscience TA AstraZeneca R&D Södertälje, Sweden; Bo Fransson, MD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, C2-84, Karolinska University Hospital Huddinge, Stockholm, Sweden
Locations (1):
- Research Site, Stockholm, Sweden